CLINICAL TRIAL: NCT04365075
Title: Excimer Laser Combined With DCB Compared With Angioplasty Alone in the Treatment of Infrapopliteal Lesions in Patients With Critical Limb Ischemia.
Brief Title: Excimer Laser Combined With DCB Compared With Angioplasty Alone in the Treatment of Infrapopliteal Lesions.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XuanwuH202001
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Critical Limb Ischemia; Infrapopliteal Lesions
Keywords: Excimer Laser; Angioplasty; drug-coated baloons
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Angioplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Excimer Laser Combined with DCB (Experimental): Using excimer laser combined with drug-coated baloons to treat infrapopliteal lesions in patients with critical limb ischemia.
  Interventions: Device: Excimer Laser Combined with DCB
- Angioplasty Alone (Active Comparator): Using angioplasty alone to treat infrapopliteal lesions in patients with critical limb ischemia.
  Interventions: Device: Angioplasty Alone

INTERVENTIONS:
Device: Excimer Laser Combined with DCB — Using excimer laser combined with drug-coated baloons to treat infrapopliteal lesions in patients with critical limb ischemia.
  Arms: Excimer Laser Combined with DCB
Device: Angioplasty Alone — Using angioplasty alone to treat infrapopliteal lesions in patients with critical limb ischemia.
  Arms: Angioplasty Alone

SUMMARY:
This study was designed to compare excimer laser combined with drug-coated baloons with angioplasty alone in the treatment of infrapopliteal lesions in patients with critical limb ischemia.

DETAILED DESCRIPTION:
This is a randomized study comparing excimer laser combined with drug-coated baloons with angioplasty alone in the treatment of infrapopliteal lesions in patients with critical limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

* The treatment vessel is DeNovo
* Stenotic (>50%) or occlusive atherosclerotic disease of infrapopliteal artery(s)
* Reference target vessel diameter between 2-4.0 mm by visual assessment
* Documented Rutherford Class 4 or 5 symptomatic critical limb ischemia
* The patient must be >18 years of age
* Life-expectancy of more than 12 months
* The patient has no child bearing potential or negative serum pregnancy test
* within 7 days of the index procedure
* The patient must be willing and able to return to the appropriate follow-up times for the duration of the study
* The patient must provide written patient informed consent that is approved by the ethics committee

Anatomic Inclusion Criteria:

* All inflow lesions successfully (<30 residual stenosis) treated prior to target lesion treatment during same procedure or according standard of care without unresolved complications
* At least one angiographically visible target at the ankle for establishment of straight line flow.

Exclusion Criteria:

* Patient refusing treatment
* The target vessel segment diameter is not suitable for available catheter design.
* Unsuccessfully treated endovascular or bypass( >30% residual stenosis) proximal ( iliac, superficial femoral, popliteal) inflow limiting arterial/graft stenosis
* Lesion lies within or adjacent to an aneurysm
* The patient has a known allergy to heparin, Aspirin or other antiaggregant therapies or a bleeding diatheses or is unable, or unwilling, to tolerate such therapies.
* The patient has a history of prior life-threatening contrast media reaction.
* The patient is currently enrolled in another investigational device or drug trial.
* The patient is currently breast-feeding, pregnant or intends to become pregnant.
* The patient is unable to provide informed consent
* The patient has end stage renal disease (currently on any form of dialysis)
* Known Left Ventricular Ejection Fraction < 35%
* The patient has had a myocardial ischemia within 30 days prior to enrollment
* The patient has had a cardiovascular accident within 90 days prior to enrollment
* Serum Creatinine > 150 µmol
* The patient has a previous bypass in the target limb
* The patient has a current systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Target lesion revascularization rate | 6-months
  Free target vascular occlusion and clinically driven target lesion revascularization rate confirmed by ultrasound examination.

SECONDARY OUTCOMES:
Incidence of major adverse events | 6-months
  Incidence of major adverse events (including operative-related arterial dissection, perforation, rupture, embolization, acute thrombosis, pseudoaneurysm, and hematoma formation).
Major amputation rate | 6-months
  The rate of major amputation.
Mortality | 6-months
  The ratio of deaths
Ankle Brachial Index | 6-months
transcutaneous oxygen pressure | 6-months
Wound healing wagner score (for patients with Rutherford classification 5) | 6-months
  Wound healing wagner score (for patients with Rutherford classification 5).
Length of hospital stay | 6-months
hospitalization costs | 6-months

CONTACTS AND LOCATIONS:
Locations (1):
- Yongquan Gu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No